CLINICAL TRIAL: NCT06297733
Title: Turkish Adaptation, Validity and Reliability of the Approaches and Study Skills Inventory in Physiotherapy Students
Status: Completed | Type: Observational
Sponsor: Istanbul Bilgi University (Other)
Responsible Party: Principal Investigator, Furkan Çakır, Principal Investigator, Istanbul Bilgi University
Other Study IDs: IstanbulBUFC3
Record Dates: First submitted 2024-02-29; First posted 2024-03-07 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Health Education
Keywords: study skills; study approaches; reliability; validity
MeSH Terms: conditions — Health Education | interventions — Reproducibility of Results

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Physiotherapy Students: The population of the research consists of undergraduate students of the physiotherapy and rehabilitation department.
  Interventions: Other: Translating the Questionnaire into Turkish and Related Processes; Other: Validity; Other: Reliability

INTERVENTIONS:
Other: Translating the Questionnaire into Turkish and Related Processes — The first step is the translation from the original language to the other language. The ideal target in the translation phase is to use people who are familiar with the structure of the original language and who are familiar with the language. Two forward translation and one reverse translation methods will be applied after obtaining the written permission of the authors. After the completion of this phase, the terminological differences arising from the translators in the translation process from the original language to Turkish will be collected and discussed on the questions. The cultural adaptation study will be terminated by determining the equivalence between the Turkish version of the inventory and the English original. The final version of the questionnaire and the necessary changes will be arranged specific to the investigator's society and the authors of the original questionnaire will be consulted and the questionnaire will be finalized.
Other: Validity — The inventory will be applied by face-to-face technique and convergent validity will be evaluated. Construct validity will be evaluated through exploratory and confirmatory factor analysis. Coefficients of fit will be calculated.
Other: Reliability — The reliability of the items will be tested with Cronbach alpha. Test-retest reliability will be measured by ICC.

SUMMARY:
The quality and quantity of learning are determined by the learning approach adopted by the student. When learning and studying approaches are mentioned, individual differences between learners' learning intentions during a learning situation or while studying and what types of strategies are used to achieve these intentions come to mind. These learning approaches are thought to determine the quality of learning outcomes. Many measurement tools have been developed to quantitatively measure learning and studying approaches. These developed tools are mostly applied at the higher education level. Among the purposes of using measurement tools; These include identifying low-performing students through screening, evaluating and identifying areas of difficulty that require prediction or improvement plans, evaluating before and after academic improvement programs, and raising awareness and advising students on their academic strengths and weaknesses.

When multidimensional measurement tools that evaluate students' study approaches and skills are examined, it is seen that the use of the Approaches and Study Skills Inventory for Students (ASSIST) tool has become widespread in recent years. This vehicle; It has been reported that it measures learning strategies and skills for different students and is sensitive enough to distinguish between learning types.

The Portuguese, Norwegian and Danish versions of the survey, which was developed in English and intended to be translated into Turkish as the Study Skills and Approaches Scale, have also been translated, its psychometric properties have been demonstrated and it has been observed that it is becoming widespread in the literature.

DETAILED DESCRIPTION:
The quality and quantity of learning are determined by the learning approach adopted by the student. When learning and studying approaches are mentioned, individual differences between learners' learning intentions during a learning situation or while studying and what kind of strategies are used to achieve these intentions come to mind. Many measurement tools have been developed to quantitatively measure learning and studying approaches. These developed tools are mostly applied at the higher education level. Among the purposes of using measurement tools; These include identifying low-performing students through screening, evaluating and identifying areas of difficulty that require prediction or improvement plans, evaluating before and after academic improvement programs, and raising awareness and advising students on their academic strengths and weaknesses.

When multidimensional measurement tools that evaluate students' study approaches and skills are examined, it is seen that the use of the Approaches and Study Skills Inventory for Students (ASSIST) tool has become widespread in recent years. This vehicle; It has been reported that it measures learning strategies and skills for different students and is sensitive enough to distinguish between learning types.

The Portuguese, Norwegian and Danish versions of the survey, which was developed in English and intended to be translated into Turkish as the Study Skills and Approaches Scale, have also been translated, its psychometric properties have been demonstrated and it has been observed that it is becoming widespread in the literature.

It is aimed to ensure the validity and reliability of this tool, which evaluates superficial, deep and strategic learning approaches on students in various undergraduate departments, and to use it as an objective scale.

The first comprehensive ASSIST assessment tool was first developed in 1998 and was structured as 64 items and 16 subheadings. The first and third sections of the form are small subsections in which the individual describes his or her learning and indicates learning preferences regarding different course types. The second part of the form, which distinguishes learning types and constitutes the focus of this study, took its final form as a 52-item, 5-point Likert form and three factors were identified as its psychometric properties were examined over time (Tait et al., 1998).

It is scored as 5=strongly agree, 4=agree, 3=not sure, 2=disagree, 1=strongly disagree. There are no reverse coded items.

There are 20 items assessing deep learning, 16 items measuring surface learning, and 16 items measuring strategic learning. Items measuring learning types are in mixed order.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-30
* Being a student at the Department of Physiotherapy and Rehabilitation of the Faculty of Health Sciences

Exclusion Criteria:

* People with vision problems that would prevent participation in the study
* Participants who have not filled out the forms completely will be excluded from the research.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The population of the research consists of undergraduate students of the physiotherapy and rehabilitation department.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Approaches and Study Skills Inventory for Students | Baseline
  Approaches and Study Skills Inventory for Students, developed by Tait et al. in 1998, is a 52-item survey that evaluates the learning behaviors of higher education students under the subheadings of deep, superficial and strategic learning. For each item, the participant is asked to mark the option that he/she thinks corresponds to the appropriate option between 0=strongly disagree and 5=strongly agree. Deep learning (article 4-7-9-11-13-17-20-21-23-26-30-33-34-36-39-43-46-47-49-52), surface learning (article 3). -6-8-12-16-19-22-25-29-32-35-38-42-45-48-51), and strategic learning (article 1-2-5-10-14-15-18 -24-27-28-31-37-40-41-44-50). There is no reverse coded item. For the original version of the form, the deep learning score varies between 0-100, and the superficial and strategic learning score varies between 0-80. The short version of the 18-item form selected from the 52-item form will also be examined.
Participant Information Form | Baseline
  Participating students will be asked for a nickname they choose, their gender, age, whether they are a physiotherapy and rehabilitation student, what grade they are in, and their current GPA score.

CONTACTS AND LOCATIONS:
Overall Officials: Ilksan Demirbuken, Prof, Study Director — Marmara University; Mine Gulden Polat, Prof, Study Director — Marmara University
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided